CLINICAL TRIAL: NCT03817918
Title: A Pilot Study of a New Ultrasonographic Tool to Assess Regional Pulmonary Strain in Patients Under General Anesthesia Using One-lung Ventilation.
Brief Title: A New Ultrasonographic Tool to Assess Pulmonary Strain in Patients Under One-lung Ventilation.
Acronym: STRAIN-VUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18.304
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Ventilator-Induced Lung Injury; Mechanical Ventilation Complication
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of local pleural strain (Experimental): The local pleural strain will be determined over three consecutive respiratory cycles using lung ultrasonography
  Interventions: Procedure: Lung ultrasonography

INTERVENTIONS:
Procedure: Lung ultrasonography — Patients undergoing thoracic surgery under general anesthesia using one-lung ventilation will have lung ultrasonography at 2 predetermined sites at four different time points

SUMMARY:
Mechanical ventilation is frequently used in the operating room and the intensive care settings. Although essential in many cases, mechanical ventilation can be responsible for ventilator-induced lung injury (VILI). The relationship between mechanical ventilation and VILI has been clearly demonstrated in animals and is highly suspected in humans. The putative mechanism responsible for VILI is excessive pulmonary strain or overdistension. Frequently observed in mechanically ventilated patients, the presence of a severe pre-existing pulmonary disease can increase the risk of overdistension. The development of a tool allowing early detection of pulmonary overdistension would represent a great asset in the prevention of VILI by allowing safer adjustments of mechanical ventilation parameters. Ultrasonographic imaging is a non-radiant, non-invasive technique already available in the intensive care setting. Already used for cardiac strain measurements, ultrasonography is a promising avenue to assess pulmonary strain.

This pilot study will aim to create a small dataset of local pleural strain values assessed at predetermined pulmonary areas using ultrasound imaging in patients undergoing thoracic surgery requiring one-lung ventilation. This dataset will be used to help plan larger scale studies.

DETAILED DESCRIPTION:
At four different time points during thoracic surgery, images of the pleura of the dependent lung will be made at 2 predetermined areas. The images will be made: after induction (tidal volume of 10 mL/kg), during two-lung ventilation (tidal volume of 10 mL/kg) and during one-lung ventilation (tidal volume of 10 mL/kg and 5 mL/kg). The sites to be studied will be: the 3rd intercostal space at the mid-clavicular line (dependent lung), the 8th intercostal space at the posterior axillary line (dependent lung). Three consecutive respiratory cycles at each site will be recorded for subsequent analysis.

Lung ultrasonography will be performed by the principal investigator and a co-investigator using a Terason (Teratech Corporation, Burlington, MA) device and a 12L5 linear ultrasound probe. For each image, the probe will be oriented perpendicularly to the pleura with the pointer towards the participant's head. A depth of 4 cm will be used and adjusted in order to have the pleural line located between the center and the three-quarts of the screen. The beam's focal zone will be positioned at the level of the pleural line. A 12 MHz frequency will be used.

Using a reference ultrasonographic image, an experienced lung ultrasonographer will segment the pleura. From this image, an algorithm will define a region of interest which will be followed throughout the rest of the images of the video sequence. Thereafter, the algorithm will calculate the various components of pulmonary strain in relation to tidal volume. The principal investigator or a co-investigator will visually validate the speckle-tracking.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery in lateral position requiring one-lung ventilation

Exclusion Criteria:

* Obesity (Body Mass Index superior to 30 kg/m2)
* Emergency surgery
* Previous thoracic procedure (chest tube, thoracotomy, thoracoscopy)
* Previous participation to the study
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Feasibility of the measurement of local pleural strain using ultrasonography | At the end of the study on Day 1
  Proportion of successfully analyzed lung ultrasonographic clips

SECONDARY OUTCOMES:
Average absolute lateral deformation | At the end of the study on Day 1
  Change in percentage from baseline expiratory values
Cumulated range of absolute lateral deformation | At the end of the study on Day 1
  Change in percentage from baseline expiratory values
Average absolute lateral shift | At the end of the study on Day 1
  Change in percentage from baseline expiratory values
Cumulated range of absolute lateral shift | At the end of the study on Day 1
  Change in percentage from baseline expiratory values
Average von mises | At the end of the study on Day 1
  Change in percentage from baseline expiratory values

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No